CLINICAL TRIAL: NCT02468895
Title: MYOPROSP: A Prospective Cohort Study to Identify a Stratified Approach in the Diagnosis, Treatment and Delivery of Care in Adult Idiopathic Inflammatory Myopathy
Brief Title: MYOPROSP - a Prospective Cohort Study in Myositis
Acronym: MYOPROSP
Status: Active, not recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: University of Bath (Other); University College, London (Other); Royal Victoria Infirmary (Other); King's College Hospital NHS Trust (Other); North Bristol NHS Trust (Other); University of Liverpool (Other); St. George's Hospital, London (Other); Northern Care Alliance NHS Foundation Trust (Other); Burton Hospitals NHS Foundation Trust (Other); Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other); Sandwell & West Birmingham Hospitals NHS Trust (Other); London North West Healthcare NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Hector Chinoy, Professor, University of Manchester
Other Study IDs: UoMMYO
Record Dates: First submitted 2014-12-05; First posted 2015-06-11 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Myositis; Idiopathic Inflammatory Myopathy
Keywords: Myositis; Idiopathic inflammatory myopathy; Antibodies; Genetics; Biomarkers
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — DNA RNA Peripheral blood mononuclear cells Serum Plasma Urine Muscle biopsies Other diagnostic tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Idiopathic Inflammatory Myopathy: PM, DM, sIBM, necrotizing myopathy, anti-synthetase syndrome, suspected myopathy

SUMMARY:
Adult patients with suspected or confirmed idiopathic inflammatory myopathy (IIM) will be recruited. Patients will be approached, consented, have baseline demographics, diagnostics and disease activity measures recorded, and blood taken. The collection of data and biological material will mirror usual clinical practice as far as possible. Subjects will ideally attend further visits at 3, 6 and 12 months to have bloods taken, outcome measures recorded and questionnaires completed.

In addition, blood, muscle biopsies and imaging undertaken as part of usual care will also be collected for research purposes to measure a number of biomarkers for the assessment of diagnostic accuracy and clinical utility evaluation. As per usual practice, a muscle biopsy will be performed at baseline, and a further biopsy offered at 6 months to assess treatment response. A magnetic resonance (MR) muscle protocol will also be performed as per usual clinical practice, and a gadolinium-enhanced MR heart scan offered. Both these scans will be repeated at 6 months. An existing electronic database entry system will be used for data entry and capture on an anonymised basis.

The study will thus be based around diagnostic evaluations and outcome measures to improve quality of care in IIM.

DETAILED DESCRIPTION:
The bioresource from this protocol, ethics application and future funding will comprise the following:

i) UKMYONET cross-sectional study ii) MYOPROSP inception cohort study iii) MYOACT novel therapies registry iv) UK neuromuscular biobank

Primary endpoint The primary study endpoint will be sensitivity to change of the biomarkers of interest.

Secondary endpoints

This will include but not limited to:

* Response to treatment
* Drug reductions and cessations due to treatment failure, adverse events and clinical remission
* Differentiation of myositis subgroups using newer imaging modalities
* Sensitivity of biomarkers to diagnose extramuscular manifestations (including myocardial and pulmonary lung disease) and predict their severity and clinical course
* Identification of novel genetic variants associated with IIM and subtypes
* Cost economic analysis
* Validations of definition of improvement criteria

Cases will be adults >18 years, with a number of different IIM clinical phenotypes encountered in clinically practice. It is vitally important that patients with suspected, but not confirmed, IIM are also included so that the natural history and subsequent final diagnoses can be tracked. Subsequent investigations will often confirm a diagnosis that was not confirmed at initial presentation. Patients who do have confirmed PM/DM will have IIM according to the Bohan and Peter criteria, which remains the internationally accepted criteria for inclusion into clinical trials. Disease duration from onset of initial symptoms would ideally be less than one year to enrich the cohort with patients of high disease activity and minimal established disease-related damage.

Patients with suspected "possible" polymyositis (PM)/dermatomyositis (DM), where a diagnosis of IIM is suspected but not confirmed probable/definite by the Bohan and Peter criteria, will also be eligible. Patients with myositis as their primary condition and also fulfilling criteria for an associated connective tissue disease, including but not limited to, systemic sclerosis, Sjogren's, SLE, rheumatoid arthritis, will also be allowed for inclusion into the study. Patients will also be eligible if they present with ILD/Raynaud's or other CTD features in association with a myositis specific antibody other than an anti-synthetase and no other obvious IIM-diagnostic features. Patients with IBM will also be accepted on to the study, meeting the revised MRC Neuromuscular criteria.

Patients will also be accepted on to the study if they possess amyopathic or hypomyopathic DM, as per the Sontheimer criteria, which states that "amyopathic DM is a subset of DM characterized by biopsy-confirmed hallmark cutaneous manifestations of classic DM occurring for 6 months or longer with no clinical evidence of proximal muscle weakness and no serum muscle enzyme abnormalities. If more extensive muscle testing is carried out, the results should be within normal limits".

STUDY METHODS:

Initial approach Patients will be sent a letter from their consultants. The letter will give a brief introduction to the proposed study and a patient information sheet will be included. A unique identifier would be assigned to each potential new recruit. Potential participants will be given a full explanation of the study and provided with a patient information sheet and consent form to sign, following the opportunity to ask any questions. If having been allowed sufficient time to consider their decision, and they want to participate, informed consent will then be sought. The samples will be anonymised, processed, and sent to The University of Manchester for storage and analysis. No treatment will be withheld for the purposes of this study.

Data collection i) UKMYONET cross-sectional study Baseline core data encompassing the clinical information outlined in UKMYONET will be collected. Blood for sera and plasma will also be collected. Retrospective data collection will also be allowed to interrogate how baseline characteristics may influence outcome.

ii) MYOPROSP inception cohort study Baseline core data encompassing the clinical information outlined in UKMYONET will be collected, and extended data on medication use and disease activity. As genetic material (DNA) does not change with time, it would only be necessary to obtain this at one time-point (0 months); however, epigenetic, psychological, clinical and serological factors will alter over the course of the treatment, therefore sequential samples will be taken at 3, 6 and 12 month time points for comparison. Whilst being taken as part of routine clinical practice, patients can also consent to have part of their muscle biopsy, used for research purposes, as well as a follow-up biopsy. If other tissues are being taken as part of routine clinical practice, the patient can also be consented for their use as part of research studies. Patients may also be approached for further clinical data collection at yearly intervals up to 5 years after inception.

iii) MYOACT novel therapies registry Baseline core data encompassing the clinical information outlined in UKMYONET will be collected, and extended data on medication use and disease activity. Patients will also be given the option to partake in MYOPROSP for blood collection.

iv) UK neuromuscular biobank Blood/tissue related to the underlying disease process will be collected if being taken for clinical purposes. Blood samples will be used to extracted DNA, RNA, PBMC (peripheral blood mononuclear cells), serum and plasma samples which will also be stored for use in future studies. Additionally, patients will be asked for their permission to use their anonymised clinical and demographic details in any future research projects.

Blood sampling Patients consenting to take part in the study will be asked to provide blood samples as outlined above at baseline, 3 months, 6 months and 12 months. Normally, it is routine clinical practice to assess patients at these time points. These blood tests will be taken in addition to routine tests required during these assessments. Hence, although an additional blood sample will be taken, no additional venepuncture will be required thus minimising any inconvenience for the patient. In exceptional circumstances, it may be required that a blood sample is taken at an extra visit if clinic/nurse time is not available for this routine sampling. Standard laboratory assays or ELISA will be used for measuring serum enzyme, cytokine and antibody levels.

Patient questionnaires Clinical data will be attained regarding their level of disability (Stanford Health Assessment Questionnaire) and health outcome (EQ-5D-5L). When patients attend for review at each of the time points (3/6/12 months), they will be asked to complete these questionnaires. If the diagnosis is DM, patients will be asked to fill in the dermatology life quality index (DLQI) questionnaire, and if IBM, the Inclusion Body Myositis Functional Related Scale (IBM-FRS). The blood samples and questionnaires will already be labelled with a unique identifier and returned to the Centre for Musculoskeletal Research, The University of Manchester, using a pre-paid, pre-addressed blood box for the blood and a separate pre-paid stamped addressed envelope for the documentation.

Core dataset

The core dataset will comprise the UKMYONET basic dataset questionnaire and bloods for serum and plasma. Consent will also allow for further data collection as per the MYOPROSP study if the patient is under regular follow up. The International Myositis Assessment and Clinical Studies (IMACS) Group have agreed core-set measures to assess myositis disease activity, including assessment of the following:

IMACS core measures of disease activity

1. Physician/patient global activity assessment by visual analogue scale
2. IMACS core measures of disease activity
3. Physical function
4. Muscle enzymes
5. Extraskeletal muscle disease
6. Physical impairment measured with the Stanford Health Assessment Questionnaire

Muscle tissue is the primary organ affected in myositis, but other organs may also be involved, hence the requirement to capture extraskeletal disease activity using the Myositis Intention to Treat Index (MITAX) and the Myositis Activity Assessment by Visual Analogue Scales (MYOACT). The Myositis Damage Index (MDI) assesses extent and severity of damage. MITAX, MYOACT and MDI are all physician-initiated questionnaires. Further optional information can also be collected if performed as part of a routine clinical assessment, eg information on endurance.

Clinical Data As well as the information in the Core dataset, data will be captured at baseline including demographics, clinical disease classification, data detailing confirmation of diagnosis (including muscle biopsy, electromyography, autoantibody status, MR findings) co-morbidities and therapies. Changes in therapy will be captured at subsequent visits along with IMACS core measures. For IBM, additional monitoring will be performed including but not limited to IBM functional related scale, 6 minute walk test, timed up and go, grip strength.

MR imaging As a sub-study, patients will be given the option of having MR imaging of the femur to image the thigh musculature, and gadolinium-enhanced MR imaging of the heart at months 0 and 6. It is normal clinical practice to perform an MR of the femur at baseline and follow-up, and would be considered best practice to MR image the heart. In patients where gadolinium contrast would be deemed high-risk (renal impairment, history of previous contrast reactions), this would not be offered. A protocol will be developed in conjunction with musculoskeletal radiology colleagues to standardise the methods used for MR imaging in the different participating centres.

Muscle biopsy At diagnosis, a muscle biopsy is routinely performed under local anaesthetic in a non-invasive fashion. Several samples are usually taken in one pass, and one sample will stored in a PAXgene tube for RNA expression studies. The remainder of the samples will be processed and analysed in the local clinical histopathological departments. Muscle biopsy specimens will be snap-frozen in isopentane using liquid nitrogen and stored at -80C. Protocols for muscle tissue mounting, sectioning and storage that have already been tested and optimised as part of the UK juvenile dermatomyositis research study will be used. A further biopsy will be planned and offered at 6 months post-recruitment into the study. Although this is not routine clinical practice, an important clinical question needs to be addressed about the clinical utility of repeat biopsy and whether it may quantify change in disease activity and thus allow for accurate decision-making about treatment reduction/escalation.

ELIGIBILITY:
Gender Both female and males

Age limits Patients >/= 18 years

Accept healthy volunteers No

Eligibility criteria

Inclusion Criteria:

* Polymyositis
* Dermatomyositis (including amyopathic)
* Inclusion body myositis
* Anti-synthetase syndrome
* Myositis overlapping with another connective tissue disorder
* Cancer-associated myositis
* Immune-mediated necrotising myopathy including statin-induced myositis
* Juvenile myositis persisting into adulthood
* Fasciitis including eosinophilic myofasciitis
* Vasculitis affecting muscle
* Granulomatous myositis
* Focal myositis
* Orbital myositis
* Suspected myositis under investigation
* CTD features in association with a myositis specific / associated antibody

Exclusion Criteria:

* Patients with disease duration >2 years
* Patients < 18 years
* Confirmed non-inflammatory myopathies
* Myositis secondary to alcohol or drug abuse
* Patients unwilling or unable to give consent
* Patients with poor or no venous access
* Patients where MR imaging is contraindicated (for MR substudy)

Study population description Patients referred to tertiary level UK myositis clinics

Sampling methods N/A, this is a prospective study of consecutive eligible patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Idiopathic Inflammatory Myopathy, UK based patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-10-04 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a significant change levels of diagnostic biomarkers. | 5 years
  This will depend on the specific biomarker/cytokine being measured

SECONDARY OUTCOMES:
Number of participants with a 20% improvement in myositis specific disease activity measures from baseline | 5 years
  As per the published International Myositis Assessment & Clinical Studies Group (IMACS) outcome measures of definition of improvement (http://www.niehs.nih.gov/research/resources/imacs/definitions/index.cfm)
Differences in frequency of genetic variants associated with IIM and subtypes compared to population matched controls | 5 years
  Specific identified genetic variants will be identified as part of large scale genetic studies

CONTACTS AND LOCATIONS:
Overall Officials: Hector Chinoy, PhD FRCP, Principal Investigator — The University of Manchester
Locations (1):
- The University of Manchester, Manchester, Please Select, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Core/extended dataset, SOP definitions, data access/sharing policies, data available for sharing and metadata to describe these, will be made available though the planned UKMYONET study website, meetings and presentations. Links to the results and the UKMYONET website will be available via the Euromyositis registry front page and links from local CoI websites. All data generated during this project will be made available to the scientific community through full publication in a timely fashion using open access in highest possible impact scientific journals, presentation at scientific conferences and via SC application for data access. Genotype data will be deposited and made available through a publically available repository, such as the European Bioinformatics Institute, for secure data storage.
Time Frame: Final study data and results will be available once data clean up and study analysis has been completed. Data clean up and study analysis ongoing . To be completed before the study end date, December 2030.
Access Criteria: Must be approved by the MYOPROSP steering Committee